CLINICAL TRIAL: NCT03619603
Title: Biomarkers and Associated Outcomes in Patients With Pneumonia
Brief Title: Biomarkers in Patients With Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, Clinical Professor, Chongqing Medical University
Other Study IDs: ChongqingMU3
Record Dates: First submitted 2018-07-26; First posted 2018-08-08 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, secretions and tissues.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identifying biomarkers in patients with pneumonia

DETAILED DESCRIPTION:
The aim of this study is to identify the biomarkers in patients with pneumonia. These biomarkers can distinguish community-acquired pneumonia, hospital-acquired pneumonia, severe pneumonia, bacterial infection, virus infection and fungal infection. Furthermore, these biomarkers can identify the efficacy of treatment in patients with different interventions.

ELIGIBILITY:
Inclusion Criteria: Healthy patients without any diseases -

Exclusion Criteria:Age less than 18 years

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with pneumonia
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | From diagnosis of pneumonia to discharge from hospital or up to 90 days, whichever came first
  Mortality is defined the patient died in hospital.

SECONDARY OUTCOMES:
severe pneumonia | From diagnosis of pneumonia to discharge from hospital or up to 90 days, whichever came first
  The pneumonia deteriorated and reached the criteria of severe pneumonia. Severe pneumonia was diagnosed according to the guideline published by ATS.
initial treatment failure | From diagnosis of pneumonia to discharge from hospital or up to 90 days, whichever came first
  Initial treatment failure means the patients' condition progressively deteriorated although comprehensive treatment was administrated. As a result, the treatment should be changed or the patient required admission to ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Duan, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sharement should be contact with us.